CLINICAL TRIAL: NCT04945252
Title: The Impact of School Teachers in Care Navigation and Signposting Dental Caries
Brief Title: The Impact of School Teachers in Care Navigation and Signposting Dental Caries in Primary School Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Khartoum Centre for Research and Medical Training (Other)
Responsible Party: Principal Investigator, Fadil Elamin, Doctor, Khartoum Centre for Research and Medical Training
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Khrt02
Record Dates: First submitted 2021-06-25; First posted 2021-06-30 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: Dental Caries in Children

STUDY DESIGN:
Intervention Model Description: non-randomized parallel design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Care Navigation group (Experimental): The teachers will signpost dental caries based on ICCMS visual criteria and refer to the nearest service. Annual monitoring of caries
  Interventions: Diagnostic Test: Signpost caries
- No internvention (No Intervention): Caries experience (dmft) activity monitored annually

INTERVENTIONS:
Diagnostic Test: Signpost caries — Identify carious lesion according to ICCMS visual criteria
  Other Names: signpost dental caries
  Arms: Care Navigation group

SUMMARY:
The study aims to investigate the role of school teachers in care navigation and signposting dental caries in primary school children.

DETAILED DESCRIPTION:
Dental caries is a multifactorial disease with high prevalence in children. Dental caries is a global public health problem with detrimental impact in developing countries. Despite advances in caries management and detection poorer countries continue to suffer a high burden of disease. Advances in care navigation and sign-posting concepts are increasingly being utilized in general health care to aid early diagnosis and ease the burden of disease in poorer communities. This study aims to investigate the role of primary school teachers as care navigators with regard to dental caries in children.

ELIGIBILITY:
Inclusion Criteria:

Healthy school children between the ages of 5-8 years Regular school attender Lives in the local village Co-operative

Exclusion Criteria:

* known medical history or disability
* irregular school attenders

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 307 (Actual)
Dates: Start 2016-06-19 (Actual); Primary Completion 2019-06-20 (Actual); Study Completion 2020-03-11 (Actual)

PRIMARY OUTCOMES:
untreated caries increment | 36 months
  decay component of the Index of decayed, extracted and filled teeth for the groups (deft)

SECONDARY OUTCOMES:
caries experience (deft) | 36 months
  deft index (for entire group)
caries experience for the most affected one third (SIC index) | 36 months
  SIC index (deft of the most affected one third of each group)
care index | 36 months
  proportion of filled and extracted teeth (df/deft)

CONTACTS AND LOCATIONS:
Locations (1):
- Khartoum Centre for Research and Medical Training, Khartoum, Sudan

IPD SHARING:
Plan to Share IPD: Undecided